CLINICAL TRIAL: NCT07226427
Title: A Phase 1, First-in-Human Study of MEN2501, a KIF18A Inhibitor, as Monotherapy in Participants With Platinum-Resistant Ovarian Cancer
Brief Title: A First-in-Human Study of MEN2501 in Participants With Platinum-Resistant Ovarian Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MEN2501-01
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Platinum-resistant Ovarian Cancer
Keywords: MEN2501; First-in-Human; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants enrolled in the Part B dose expansion will be randomized between expansion doses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: MEN2501 Dose Escalation (Experimental)
  Interventions: Drug: MEN2501
- Part B: MEN2501 Dose Expansion & Optimization (Experimental)
  Interventions: Drug: MEN2501

INTERVENTIONS:
Drug: MEN2501 — Oral tablet

SUMMARY:
This is a first-in-human, open-label, dose-escalation, dose-optimization trial designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and antitumor activity of MEN2501 monotherapy in adult participants with platinum-resistant ovarian cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must have a histopathologically confirmed diagnosis of high-grade serous ovarian cancer, primary peritoneal cancer, or fallopian tube cancer.

Key Exclusion Criteria:

* Participants with primary platinum-refractory disease.

Note: Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-12-02 (Estimated); Study Completion 2028-06-02 (Estimated)

PRIMARY OUTCOMES:
Part A Only: Number of Participants with Dose-limiting Toxicities (DLTs) | Cycle 1 (28 days/cycle)
Part B Only: Recommended Phase 2 Dose (RP2D) of MEN2501 | Up to approximately 6 months

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events | Up to approximately 7 months
Overall Response Rate | Up to approximately 7 months
Duration of Objective Response | Up to approximately 7 months
Clinical Benefit Rate | Up to approximately 7 months
Progression-free Survival | Up to approximately 12 months
Overall Survival | Up to approximately 12 months
Time To Response | Up to approximately 7 months
Area Under the Plasma Concentration-time Curve (AUC) of MEN2501 | Up to approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Stemline Therapeutics, Inc.
Locations (1):
- NEXT Virginia, Fairfax, Virginia, United States